CLINICAL TRIAL: NCT00827671
Title: Multi-Modality Treatment of Resectable Oesophageal Adenocarcinoma Using Peri-operative Chemotherapy With Additional Pre-operative Combined Radiotherapy and Cetuximab
Brief Title: Study of Combination of Cetuximab and Radiotherapy Added to the Standard Treatment for Oesophageal Adenocarcinoma
Acronym: TRACC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Experimental treatment not feasible due to high rate of drop out
Sponsor: P.O. Witteveen (Other)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor-Investigator, P.O. Witteveen, Head of Department, UMC Utrecht
Organization: UMC Utrecht (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL23124.041.08; 2008-002203-13 (EudraCT Number)
Record Dates: First submitted 2009-01-22; First posted 2009-01-23 (Estimated); Last update posted 2018-03-09 (Actual); Status verified 2018-03

CONDITIONS: Resectable Esophageal Cancer
MeSH Terms: interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pre-operative chemotherapy (Other)
  Interventions: Drug: cetuximab; Radiation: radiotherapy to oesophageal tumour

INTERVENTIONS:
Drug: cetuximab — cetuximab initial dose 400 mg/m2 iv 1 week before start radiotherapy and subsequent weekly doses of 250 mg/m2 iv for the duration of the radiation treatment
  Other Names: erbitux; c225
Radiation: radiotherapy to oesophageal tumour — 45 Gy delivered in 25 fractions of 1.8 Gy 5d/wk

SUMMARY:
The purpose of this study is to determine whether the addition of the combination between cetuximab and radiotherapy to the standard chemotherapy for resectable oesophageal cancer is safe and adds efficacy.

DETAILED DESCRIPTION:
This study aims at developing a novel strategy to optimize the treatment of oesophageal adenocarcinoma and gastro-oesophageal junctional tumors with curative intent. Surgery in combination with peri-operative chemotherapy, using the combination epirubicin, cisplatin and 5-FU, as defined by the recent MAGIC trial, results in 13% increase in 5-yr survival. To improve the outcome of patients with this disease we hypothesize that the addition of pre-operative combined cetuximab-radiotherapy (cetux-RT) treatment could improve the outcome of this patient category through better local control.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven resectable adenocarcinoma of the lower oesophagus and gastric-oesophageal junction
* Tumour stage: T2-3 N0-1 M0, as assessed by endoscopic ultrasound and CT-scan of thorax and abdomen and ultrasound neck region. For the patients treated in this study the gastro-oesophageal junctional tumors will be staged as oesophageal tumors with respect to their lymphnode metastases.
* Age >18y and written informed consent after at least 4 days of deliberation time from the moment the patient information has been given and has been explained.
* Weight loss < 10% in 0.5 yr
* WHO performance status 0-1
* No prior radiotherapy or chemotherapy for the adenocarcinoma of the oesophagus

Exclusion Criteria:

* Previous malignancy other than basal cell carcinoma of the skin or local resection for cervical carcinoma in situ.
* Inadequate organ function as defined by:
* Inadequate haematology (Hb < 5,5 mmol/L (red blood cell transfusions are allowed to increase the Hb at the discretion of the investigator) - neutrophils < 1,5 109/L -platelets <100*109/L),
* Liver enzyme elevation (bili > 1,5*ULN - ASAT > 2,5*ULN - ALAT > 2,5*ULN) or
* Impaired renal function (creatinine clearance by cockcroft < 60 cc/min)
* Proteinuria >1,0gr/24hr
* Tumour stage: M1a and/or tumour length > 8 cm and/or > 5 cm radially
* Major surgery within 4 weeks prior to the start of study treatment
* Bleeding disorder
* Known allergy to one of the study drugs used
* Use of any substance known to interfere with the chemotherapy clearance
* Previous radiotherapy to the chest
* Significant concomitant diseases preventing the safe administration of study drugs or likely to interfere with study assessments
* Uncontrolled angina pectoris; cardiac failure or clinically significant arrhythmias
* Continuous use of immunosuppressive agents
* Concurrent use of the antiviral agent sorivudine or chemically related analogues, such as brivudine
* Prior exposure to anti-EGFR targeting agents.
* Hearing loss > 25 dB under normal
* Neurotoxicity > CTC grade 1
* Pregnancy or breast feeding
* Patients (M/F) with reproductive potential not implementing adequate contraceptive measures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-03 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
pathological complete remission | 1 month
  determination of tumor residual cell content in surgical specimen
Resectability rate defined as the number of patients abke to undergo resection after neo-adjuvant treatment | 6 months

SECONDARY OUTCOMES:
Adverse events during neo-adjuvant treatment as defined by NIH CTCAE v3.0 | 5 months
Complications in the post-operative period (defined as 4 weeks after surgery) that can be attributed to surgical procedures | 4 weeks
Progression free survival and overall survival | 5 years
Define local (locoregional lymphnode metastasis as defined by TNM classification/ malignant peritonitis/ solid masses within the anatomic region of the esophagus) vs distant metastases as first manifestation of recurrence | 5 years
The number of R0 resection determined by the pathologist | after surgery

CONTACTS AND LOCATIONS:
Overall Officials: M. P. Lolkema, MD/PhD, Principal Investigator — UMC Utrecht
Locations (1):
- UMC Utrecht, Utrecht, Netherlands

REFERENCES:
- [Derived] Ubink I, van der Sluis P, Schipper M, Reerink O, Voest E, Borel-Rinkes I, Wijrdeman H, Vleggaar F, Agterof M, Overkleeft E, Siersema P, van Hillegersberg R, Lolkema MP. Adding preoperative radiotherapy plus cetuximab to perioperative chemotherapy for resectable esophageal adenocarcinoma: a single-center prospective phase II trial. Oncologist. 2014 Jan;19(1):32-3. doi: 10.1634/theoncologist.2013-0254. Epub 2013 Dec 12. PMID 24335595